CLINICAL TRIAL: NCT03332303
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multi-Site Study to Evaluate Therapeutic Equivalence of Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) to Estrace® Cream (Warner Chilcott) in Treatment of Vulvar and Vaginal Atrophy
Brief Title: Study to Evaluate the Equivalence of Estradiol Vaginal Cream to Reference Standard in the Treatment of Vaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prasco LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71759501
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-03

CONDITIONS: Vulvar and Vaginal Atrophy
Keywords: Vaginal Dryness; Vaginal and/or Vulvar Irritation/Itching; Dysuria; Vaginal Pain and Bleeding
MeSH Terms: conditions — Pruritus; Dysuria; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) (Experimental): Estradiol Vaginal Cream, USP, 0.01%, administered once daily for 7 days.
  Intervention: Drug: Estradiol Vaginal Cream, USP, 0.01%
  Interventions: Drug: Estradiol Vaginal Cream
- Active Comparator: Estrace® Cream (Active Comparator): Estrace® Cream (Estradiol Vaginal Cream, USP, 0.01%), administered once daily for 7 days.
  Intervention: Drug: Estrace® Cream (Estradiol Vaginal Cream, USP, 0.01%)
  Interventions: Drug: Estrace® Cream
- Placebo Comparator: Placebo (Test vehicle cream) Vaginal Cream (Placebo Comparator): Placebo (Test vehicle cream) Vaginal Cream, administered once daily for 7 days.
  Intervention: Drug: Placebo (Test vehicle cream) Vaginal Cream
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Estrace® Cream — Estrace® Cream
  Other Names: Estradiol Vaginal Cream
  Arms: Active Comparator: Estrace® Cream
Drug: Estradiol Vaginal Cream — Estradiol Vaginal Cream
  Arms: Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC)
Drug: Vehicle Cream — Vehicle Cream
  Other Names: Placebo
  Arms: Placebo Comparator: Placebo (Test vehicle cream) Vaginal Cream

SUMMARY:
The objectives of this study are to evaluate the therapeutic equivalence of the Test formulation, Estradiol Vaginal Cream 0.01% (Prasco, LLC) to the marketed product, Estrace® Cream (estradiol vaginal cream, 0.01%) in patients with vulvar and vaginal atrophy, and compare the safety of Test, Reference and Placebo treatments in patients with vulvar and vaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed IRB-approved informed consent form that meets all criteria of current FDA regulations.
2. Postmenopausal females aged 30-75 years inclusive. Postmenopausal is defined as follows:

   1. At least 6 months of spontaneous amenorrhea.
   2. At least 6 weeks post-surgical bilateral oophorectomy, with or without hysterectomy.
   3. Hysterectomy without oophorectomy if of age that the Investigator believes would have naturally reached 12 months of spontaneous amenorrhea if uterus had remained intact.
3. Patients with a serum Follicle Stimulating Hormone (FSH) level of ≥ 40 mIU/mL at Screening.
4. Have ≤ 5% superficial cells on vaginal smear cytology.
5. Have a vaginal pH > 5.0.
6. At least one of the following patient self-assessed moderate to severe symptoms of VVA from the following list that is identified by the patient as being the most bothersome to her:

   * Vaginal Dryness
   * Vaginal and/or Vulvar Irritation/Itching
   * Dysuria
   * Vaginal Pain associated with sexual activity
   * Vaginal Bleeding associated with sexual activity (presence or absence)

     * Provided that patient is currently sexually active and plans to remain so throughout the study.
7. Have "Normal" Screening mammogram completed within 9 months before Screening in all patients > 40 years old, with no findings that, in the opinion of the Investigator, would indicate any suspicion of breast malignancy.
8. Normal clinical breast examination at Screening.
9. Patients with an intact uterus (including patients who underwent a partial hysterectomy) must have a documented papanicolaou (PAP) smear conducted within the previous 12 months with no findings that the Investigator believes would contraindicate the use of topical vaginal estradiol.
10. Patients with an intact uterus should have vaginal ultrasonography results within 3 months before Screening to confirm an inactive endometrial lining, defined as endometrial thickness < 4 mm.

Exclusion Criteria:

1. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
2. Any clinically significant laboratory finding that, in the Investigator's opinion would contraindicate the use of estradiol or compromise patient safety.
3. Patients with known concurrent vaginal infections including but not limited to: Candida albicans, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhea or Gardnerella vaginalis.
4. Patients with active vaginal herpes simplex infection or have had an outbreak within 30 days before the Screening.
5. Patients with known, suspected or current history of carcinoma of the breast.
6. Patients with baseline systolic blood pressure of > 150 mmHg and/or diastolic pressure > 90 mmHg.
7. Any patient with past or current undiagnosed vaginal bleeding or significant risk factors for endometrial cancer.
8. Any history of estrogen-dependent neoplasia (e.g., endometrial cancer).
9. Patients with known, suspected or current history of hormone dependent tumor.
10. History of acute thrombophlebitis or thromboembolic disorder.
11. Any prescription treatment for vaginal dryness/irritation within 14 days before Screening or any over-the-counter or natural remedies within 7 days before Screening.
12. Any prescription treatment for bacterial or yeast infections within 30 days before Screening.
13. Fasting triglyceride levels > 350 mg/dL.
14. History of radiation therapy or recent (within previous 6 weeks) surgical therapy to the vaginal or cervical areas.
15. Any known or suspected allergies that, in the Investigator's opinion, would compromise the safety of the patient.
16. Patients who have used vaginal hormonal products (rings, creams, gels) within the 7 days before Screening.
17. Patients who have used transdermal estrogen and/or progestin therapy within the 28 days before Screening.
18. Patients who have used oral estrogen and/or progestin therapy or intrauterine progestin therapy within the 56 days before Screening.
19. Patients who have used progestin implants or estrogen alone injectable drug therapy within the 3 month before Screening.
20. Patients who have used estrogen pellet therapy or progestin injectable drug therapy within 6 months before Screening.
21. History of significant alcohol abuse within 1 year prior to Screening or regular use of alcohol within 6 months before Screening (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
22. History of significant drug abuse within 1 year prior to Screening, use of soft drugs (such as marijuana) within 3 months before Screening, or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year before Screening.
23. Use within 30 days of Screening with known strong CYP3A4 inducers or inhibitors that, in the opinion of the Investigator, may affect estrogen metabolism. Examples of strong CYP3A4 inhibitors are macrolide antibiotics such as clarithromycin and telithromycin; azole antifungals such as itraconazole and ketoconazole; antidepressants such as nefazodone; and foods such as grapefruit or grapefruit juice. Examples of strong CYP3A4 inducers are anticonvulsants such as carbamazepine and phenytoin; bactericidals such as rifampin and rifabutin; and natural health products such as St. John's wort.
24. Inability to understand the requirements of the study and the relative information or are unable or not willing to comply with the study protocol.
25. Receipt of any drug as part of a research study within 30 days before Screening.
26. Employees of the Investigator or research center or their immediate family members.
27. Patients who have participated in this study previously.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Gongas, Study Director — Novum
Locations (27):
- United States (27):
  - Douglas Young, MD, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Women's Health Care Research Corp., San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Avail Clinical Research, LLC, DeLand, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Health Awareness, Inc., Port Saint Lucie, Florida
  - Physician Care Clinical Research, LLC, Sarasota, Florida
  - Well Pharma Medical Research Group, South Miami, Florida
  - Meridien Research, Inc., St. Petersburg, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Praetorian Pharmaceutical, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Canton Obstetrics and Gynecology, Canton, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Women's Clinic of Lincoln, Lincoln, Nebraska
  - Lawrence Ob-Gyn Clinical Research, LLC, Lawrenceville, New Jersey
  - Aventiv Research, Inc., Columbus, Ohio
  - Novum PRS, Pittsburgh, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Vernon & Waldrep OBGYN Associates, Dallas, Texas
  - Women's Clinical Research Center dba Seattle Women's Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 540 participants were randomized at 26 investigative sites (medical clinic/research) located in the US. 215 participants were assigned to the test drug arm, 216 participants were assigned to the reference drug arm, and 109 participants were assigned to the placebo arm. The first subject was enrolled on 26-OCT-2017 and the last subject visit was 15-MAR-2018. The study duration was approximately 5 months.
Pre-assignment Details: Following the 28-day screening period, participants who continued to meet the inclusion/exclusion (I/E) criteria were randomly assigned to treatment on a 2:2:1 ratio of test Estradiol Vaginal Cream USP, 0.01%; Estrace Vaginal Cream USP, 0.01%; or Placebo test vehicle vaginal cream.
Groups:
- Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC): Estradiol Vaginal Cream, USP, 0.01%, administered once daily for 7 days.
  Intervention: Drug: Estradiol Vaginal Cream, USP, 0.01%
  Estradiol Vaginal Cream: Estradiol Vaginal Cream
- Active Comparator: Estrace® Cream: Estrace® Cream (Estradiol Vaginal Cream, USP, 0.01%), administered once daily for 7 days.
  Intervention: Drug: Estrace® Cream (Estradiol Vaginal Cream, USP, 0.01%)
  Estrace® Cream: Estrace® Cream
- Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream: Placebo (Test vehicle cream) Vaginal Cream, administered once daily for 7 days.
  Intervention: Drug: Placebo (Test vehicle cream) Vaginal Cream
  Vehicle Cream: Vehicle Cream
Period: Overall Study
Arm/Group | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) | Active Comparator: Estrace® Cream | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream
Started | 215 | 216 | 109
Safety Population (All participants who were randomized and received study product.) | 215 | 216 | 109
Modified Intention to Treat (mITT) Population (mITT = All participants administered at least one dose of randomized study product and had a post-randomization evaluation.) | 214 | 213 | 109
Per Protocol (PP) Population (PP = All participants who met all I/E criteria, had no significant protocol deviations, did not develop concurrent vaginal infection, completed Day 8 or Day 9 visit, and administered 75% - 125% of required doses.) | 196 | 196 | 104
Completed | 196 | 196 | 104
Not Completed | 19 | 20 | 5
Not completed — Participant did not dose | 1 | 2 | 0
Not completed — Participant did not have at least one post-randomization evaluation | 0 | 1 | 0
Not completed — Participant developed concurrent vaginal infection/illness | 4 | 1 | 0
Not completed — Participant did not administer 75-125% of intended dose | 0 | 3 | 0
Not completed — Participant did not complete Study Visit 3 within Day 8 - Day 9 window | 10 | 10 | 3
Not completed — Participant did not meet all inclusion/exclusion criteria | 4 | 2 | 2
Not completed — Participant had a significant protocol deviation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and administered at least 1 dose of study drug (Safety Population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) | Active Comparator: Estrace® Cream | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream | Total
Number analyzed (Participants) | 215 | 216 | 109 | 540
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (5.5) | 60.7 (6.2) | 61.2 (6.1) | 61.0 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 216 | 109 | 540
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 34 | 23 | 91
  Not Hispanic or Latino | 181 | 182 | 86 | 449
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 25 | 28 | 9 | 62
  White | 185 | 182 | 99 | 466
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 215 | 216 | 109 | 540
Natural or Surgical Menopause [Count of Participants; unit: Participants]
  Natural Menopause | 154 | 141 | 78 | 373
  Surgical Menopause | 61 | 75 | 31 | 167
Vaginal Dryness [Count of Participants; unit: Participants]
  None | 0 | 3 | 1 | 4
  Mild | 7 | 6 | 3 | 16
  Moderate | 127 | 114 | 53 | 294
  Severe | 81 | 93 | 52 | 226
Vaginal/Vulvar Irritation/Itching [Count of Participants; unit: Participants]
  None | 107 | 104 | 48 | 259
  Mild | 53 | 49 | 27 | 129
  Moderate | 45 | 54 | 28 | 127
  Severe | 10 | 9 | 6 | 25
Dysuria [Count of Participants; unit: Participants]
  None | 173 | 174 | 77 | 424
  Mild | 30 | 29 | 21 | 80
  Moderate | 10 | 12 | 9 | 31
  Severe | 2 | 1 | 2 | 5
Vaginal Pain During Sexual Activity [Count of Participants; unit: Participants]
  None | 12 | 9 | 4 | 25
  Mild | 11 | 6 | 11 | 28
  Moderate | 59 | 69 | 22 | 150
  Severe | 81 | 83 | 49 | 213
  Not Reported | 52 | 49 | 23 | 124
Vaginal Bleeding During or After Sexual Activity [Count of Participants; unit: Participants]
  Absent | 131 | 136 | 67 | 334
  Present | 32 | 31 | 19 | 82
  Not Reported | 52 | 49 | 23 | 124
Most Bothersome Sign or Symptom [Count of Participants; unit: Participants]
  Vaginal Dryness | 130 | 131 | 63 | 324
  Vaginal/Vulvar Irritation/Itching | 13 | 14 | 9 | 36
  Dysuria | 1 | 1 | 0 | 2
  Vaginal Pain during Sexual Activity | 71 | 70 | 37 | 178
  Vaginal Bleeding during or after Sexual Activity | 0 | 0 | 0 | 0
% of Basal/Parabasal Cells [Mean (Standard Deviation); unit: percent] — Population: All participants who were randomized and administered at least 1 dose of study drug (Safety Population) and with evaluable basal/parabasal cells data.
  percent
    number analyzed (Participants) | 214 | 215 | 109 | 538
    (all) | 41.6 (36.1) | 36.0 (36.9) | 39.3 (36.0) | 38.9 (36.4)
% of Intermediate Cells [Mean (Standard Deviation); unit: percent] — Population: All participants who were randomized and administered at least 1 dose of study drug (Safety Population) and with evaluable intermediate cells data.
  percent
    number analyzed (Participants) | 214 | 215 | 109 | 538
    (all) | 57.4 (35.5) | 62.8 (36.3) | 59.5 (35.4) | 62.7 (34.8)
% of Superficial Cells [Mean (Standard Deviation); unit: percent] — Population: All participants who were randomized and administered at least 1 dose of study drug (Safety Population) and with evaluable superficial cells data.
  percent
    number analyzed (Participants) | 214 | 215 | 109 | 538
    (all) | 1.1 (1.5) | 1.1 (1.6) | 1.2 (1.4) | 1.1 (1.5)
Vaginal pH [Mean (Standard Deviation); unit: pH] | 6.2 (0.7) | 6.2 (0.7) | 6.2 (0.7) | 6.2 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint
Description: The primary efficacy endpoint is the number of participants in each treatment group that were identified as Responders at the end of the treatment period evaluated on Day 8 or Day 9. A Responder was defined as a participant with at least a 25% reduction from baseline in the sum of % basal/parabasal + % intermediate cells on vaginal cytology AND vaginal pH < 5.0 with a change from baseline vaginal pH of at least 0.5. Any participant who withdrew from the study because of lack of efficacy was included as a non-responder.
Time Frame: Study Day 8 or Study Day 9
Population: Therapeutic Equivalence Between Experimental and Active Comparator Arms: Per Protocol (PP) Population Superiority over Placebo: Modified Intent-to-treat population (mITT, all randomized study participants who administered at least one dose of randomized study product and had a post-randomization evaluation)
Measure: Number; unit: participants
Arm/Group | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) | Active Comparator: Estrace® Cream | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream
Number analyzed (Participants) | 214 | 213 | 109
participants
  Equivalence: PP Population: number analyzed (Participants) | 196 | 196 | 0
  Equivalence: PP Population | 49 | 59 |
  Superiority: mITT Population | 52 | 63 | 1
Statistical Analysis 1: Comparison: Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) vs Active Comparator: Estrace® Cream; Therapeutic equivalence was evaluated for both primary and secondary endpoints in the per-protocol (PP) population; Test type: Equivalence — If the 90% confidence interval (calculated using Yates' continuity correction) on the absolute difference between the proportion of patients identified as Responders in the Test and Reference groups (pT - pR) is contained within the range [-20%, +20%] then therapeutic equivalence of the Test product to the Reference product was considered to have been demonstrated; Mean Difference (Final Values) = -5.1, 90% CI 2-sided [-13.0 to 2.8]
Statistical Analysis 2: Comparison: Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) vs Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream; Superiority of the Test and Reference products against the Placebo product for the primary endpoint was evaluated in the modified Intent-to-Treat (mITT) population using last observation carried forward (LOCF); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance is p < 0.05; % Difference = 23.4
Statistical Analysis 3: Comparison: Active Comparator: Estrace® Cream vs Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance is p < 0.05; % Difference = 28.7

2. Secondary Outcome: The Secondary Efficacy Endpoint
Description: The secondary efficacy endpoint is the number of participants in each treatment group that are considered a Treatment Success at the end of the treatment period evaluated on Day 8 or Day 9. A "Treatment Success" is defined as a score of 0 or 1 on Day 8 or Day 9 for the symptom identified at baseline as the most bothersome. This evaluation will be based on (one) participant self-assessed symptom of VVA (vaginal dryness, vaginal and/or vulvar irritation/itching, dysuria, or vaginal pain associated with sexual activity) on a scale of 0 to 3 where 0 = none and 3 = severe. Evaluation of vaginal bleeding during sexual activity will be based on a score of 1 (presence) if it is identified by the participant as the most bothersome symptom at baseline and a score of 0 (absent) on Day 8 or Day 9.
Time Frame: Study Day 8 or Study Day 9
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) | Active Comparator: Estrace® Cream | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream
Number analyzed (Participants) | 214 | 213 | 109
participants
  Equivalence: PP Population: number analyzed (Participants) | 196 | 196 | 0
  Equivalence: PP Population | 112 | 116 |
  Superiority: mITT Population | 122 | 127 | 63
Statistical Analysis 1: Comparison: Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) vs Active Comparator: Estrace® Cream; Therapeutic equivalence was evaluated for both primary and secondary endpoints in the per-protocol (PP) population; Test type: Equivalence — If the 90% confidence interval (calculated using Yates' continuity correction) on the absolute difference between the proportion of patients identified as Treatment Successes in the Test and Reference groups (pT - pR) is contained within the range [-20%, +20%] then therapeutic equivalence of the Test product to the Reference product was considered to have been demonstrated; Mean Difference (Final Values) = -2.0, 90% CI 2-sided [-10.7 to 6.7]
Statistical Analysis 2: Comparison: Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) vs Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream; Superiority of the Test and Reference products against the Placebo product for the secondary endpoint was evaluated in the modified Intent-to-Treat (mITT) population using last observation carried forward (LOCF); Test type: Superiority — To conclude superiority of the Test product over Placebo, the proportion of Treatment Successes in the Test product group must be numerically and statistically superior to that of the Placebo (p < 0.05; using a two-sided Cochran-Mantel-Haenszel [CMH] test); p = 0.8068, Cochran-Mantel-Haenszel; % Difference = -0.8
Statistical Analysis 3: Comparison: Active Comparator: Estrace® Cream vs Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream; [analysis description as in outcome 2, analysis 2]; Test type: Superiority — To conclude superiority of the Reference product over Placebo, the proportion of Treatment Successes in the Reference product group must be numerically and statistically superior to that of the Placebo (p < 0.05; using a two-sided Cochran-Mantel-Haenszel [CMH] test); p = 0.8003, Cochran-Mantel-Haenszel; % Difference = 1.8

3. Other Pre Specified Outcome: Duration of Post-menopausal Status (Years)
Description: Baseline Characteristic for Participants who reported Natural Cause for Menopause (Total n = 373 patients) with mean and standard deviation (SD) evaluated per Arm/Group at Visit 1 (Day -28 to Day -1) during Medical History and Demographics Screening
Time Frame: Visit 1 (Day - 28 to Day -1)
Population: Participants who reported Natural Cause for Menopause during Medical History and Demographics Screening
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) | Active Comparator: Estrace® Cream | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream
Number analyzed (Participants) | 154 | 141 | 78
years | 11.1 (6.4) | 11.4 (6.5) | 12.3 (7.6)

ADVERSE EVENTS:
Time Frame: 8 or 9 Days (Visit 2 [Day 1; Randomization] to Visit 3 [Day 8 or Day 9])
Arm/Group | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) | Active Comparator: Estrace® Cream | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/216 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/215 | 1/216 | 0/109
Other Adverse Events (participants affected / at risk) | 66/215 | 59/216 | 23/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) (N=215) | Active Comparator: Estrace® Cream (N=216) | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream (N=109)
Exacerbation of Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — SAE required hospitalization, but was determined not to be related to the study product and no action was taken regarding the study product.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Estradiol Vaginal Cream, USP, 0.01% (Prasco LLC) (N=215) | Active Comparator: Estrace® Cream (N=216) | Placebo Comparator: Placebo (Test Vehicle Cream) Vaginal Cream (N=109)
Vertigo Positional (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distention (Gastrointestinal disorders) | 6 | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 7 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Vulvitis (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 3 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 1 | 0 | 0
Smear vaginal abnormal (Investigations) | 5 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 5 | 3
Hyperaesthesia (Nervous system disorders) | 0 | 3 | 0
Migraine (Nervous system disorders) | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 3 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 0 | 1 | 0
Breast discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 1
Breast tenderness (Reproductive system and breast disorders) | 5 | 6 | 1
Genital erosion (Reproductive system and breast disorders) | 0 | 0 | 1
Genital paresthesia (Reproductive system and breast disorders) | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 2 | 4 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 7 | 5 | 2
Uterine spasm (Reproductive system and breast disorders) | 1 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal dysplasia (Reproductive system and breast disorders) | 2 | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vulval edema (Reproductive system and breast disorders) | 1 | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 5 | 2 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 2 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 2 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 6 | 3 | 0
Vulvovaginal swelling (Reproductive system and breast disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03332303/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT03332303/SAP_003.pdf